CLINICAL TRIAL: NCT06955884
Title: Patient Experience of Transoral Versus Transnasal Awake Tracheal Intubation With Flexible Bronchoscopy - an Observational Study
Brief Title: Patient Experience of Transoral Versus Transnasal Awake Tracheal Intubation
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-101503-BO-ff
Record Dates: First submitted 2025-04-22; First posted 2025-05-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Airway Management; Fiberoptic Guided Intubation; Patient Experience
Keywords: airway management; flexible endoscopy guided intubation; patient discomfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transnasal ATI:FB: Patients undergoing airway management via the transnasal route
- Transoral ATI:FB: Patients undergoing airway management via the transoral route

SUMMARY:
Airway management problems are key drivers for anesthesia-related adverse events. Awake tracheal intubation using flexible bronchoscopy and preserved spontaneous breathing (ATI:FB) is a recommended technique to manage difficult tracheal intubation in anaesthesia, intensive care and emergency medicine. ATI:FB is regarded as the gold standard of tracheal intubation in many scenarios, however there is insufficient data on the patients experience while undergoing this form of airway management. ATI:FB can be facilitated using either a transnasal or transoral route. The study aims to compare patient-centred and operator-focused outcome parameters between these two different approaches with a focus on patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for surgery requiring tracheal intubation
* patients with an anticipated difficult airway requiring ATI:FB
* consent by the patient
* minimum 18 years of age

Exclusion Criteria:

* patients scheduled for surgery requiring tracheal intubation
* patients not scheduled for ATI:FB
* pregnant or breastfeeding patients
* consent withheld or not possible to obtain by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery requiring general anaesthesia at the study center university hospital medical center
Sampling Method: Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Patient reported discomfort experienced during ATI:FB | 24 hours after anaesthesia
  recorded on a visual analog scale (1-100; lower values better)

SECONDARY OUTCOMES:
Patient reported recall of the ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported pain experienced during ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported fear experienced during ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported feeling of suffocation experienced during ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported dyspnea experienced during ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported distress experienced during ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported coughing experienced after ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported dry throat experienced after ATI:FB? | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported hoarseness experienced after ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported sleeping problems experienced after ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported occurrence of nightmares experienced after ATI:FB | 24 hours after airway management
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported preoperative expectation of discomfort to be experienced during ATI:FB | during preoperative assessment
  yes/no and on a visual analog scale (1-100; lower values better)
Patient reported preoperative fear of airway management | during preoperative assessment
  yes/no and on a visual analog scale (1-100; lower values better)
First attempt success | 1 hour
  number of participants with successful ATI:FB with only one attempt
Number of bronchoscopy attempts | 1 hour
  Observed during airway management
Number of intubation attempts | 1 hour
  Observed during airway management
Successful ATI:FB | 1 hour
  Number of participants with successful ATI:FB
Successful bronchoscopy | 1 hour
  Number of participants with successful bronchoscopy
Successful tube placement | 1 hour
  Number of participants with successful tracheal tube placement
Conversion from transnasal to transoral bronchoscopy or vice versa | 1 hour
  Observed during airway management
Conversion to another type of airway management | 1 hour
  Observed during airway management
Percentage of glottic opening | 1 hour
  Grading of the best view obtained during laryngoscopy (%)
Glottic view | 1 hour
  Grading of the best view obtained using landmarks (6 stages)
Time to best glottic view | 1 hour
  Recorded during airway management
Time to intubation | 1 hour
  Recorded during airway management
Lowest oxygen saturation | 1 hour
  Measured during airway management (%)
Endtidal CO2 | 1 hour
  First value measured after intubation in mmHg
Airway obstructions requiring external manipulation | 1 hour
  yes/no
Hypoxia | 1 hour
  Lowest peripheral oxygen saturation measured by pulsoximetry in %
Cardiovascular event requiring intervention (hypotension/bradycardia) | 1 hour
  Observed during airway management
Cardiovascular event requiring intervention (hypertension, tachycardia) | 1 hour
  Observed during airway management
Additional manoeuvres and adjuncts | 1 hour
  Observed during airway management
Airway-related complications | 1 hour
  Recorded during airway management
Anaesthesia alert card issue | 1 hour
  Recorded after airway management
Recommendation for future airway management | 1 hour
  Recorded after airway management
Richmond Agitation-Sedation Scale | 1 hour
  Observed during airway management (-5 to 4; lower values indicate deeper sedation)
Subjective reporting of difficulty of sedation, topicalisation, bronchoscopy and tube placement | 1 hour
  On a visual analog scale (1-100)
Preparation time | 1 hour
  Recorded during airway management

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No